CLINICAL TRIAL: NCT07123012
Title: RELATIONSHIP OF REDUCED HAMSTRING FLEXIBILITY WITH LUMBOPELVIC RHYTHM AND MUSCLE ACTIVATION: A CROSS-SECTIONAL BIOMECHANICAL ANALYSIS
Brief Title: RELATIONSHIP OF REDUCED HAMSTRING FLEXIBILITY WITH LUMBOPELVIC RHYTHM AND MUSCLE ACTIVATION
Acronym: RELHAM
Status: Completed | Type: Observational
Sponsor: Sahmyook University (Other)
Responsible Party: Sponsor
Other Study IDs: SYU 2025-03-033-002
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hip Functional Restriction; Lumbar Spine Biomechanics; Lumbar Muscle Activation
Keywords: hamstring muscles; Lumbar vertabrae; Pelvis; Electromyography; Range of Motion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Short: Individuals with an SLR of 60 ° or less
- Normal: Individuals with an SLR between 60 ° and 80 °
- Normal long: Individuals with an SLR of more than 80 °

SUMMARY:
Key Findings (narrative form) The study examined how hamstring flexibility influences the way the lumbar spine and pelvis share movement during forward bending and how this affects muscle activity.

1. Flexibility and lumbar contribution When participants had tighter hamstrings, their lower back took on a larger share of the bending motion. In the full forward-bend task this relationship was strong, while in the partial bend it was still clearly evident. In other words, limited hamstring length forces the spine to bend more to reach the same position.
2. Meaningful flexibility thresholds

   Participants were divided into three straight-leg-raise (SLR) groups:
   * ≤ 60 ° (short hamstrings)
   * 61-79 ° (moderate flexibility)
   * ≥ 80 ° (good flexibility) Those in the ≤ 60 ° group showed a significantly higher lumbar contribution in both bending tasks than their more flexible peers. Once SLR exceeded roughly 60 °, additional gains in flexibility produced only modest further improvement in spine-pelvis balance, suggesting that 60 ° is a clinically important threshold.
3. When the differences appear The greatest gap between flexibility groups occurred during the first half of the bend-particularly as participants began to lean forward. As they returned to upright, the differences narrowed. This indicates that early-phase movement is the critical moment when tight hamstrings shift load onto the lumbar spine.
4. Impact on muscle activity Better hamstring flexibility was linked to a more even distribution of work between the lumbar extensor muscles and the hamstrings themselves. Participants with looser hamstrings did not have to activate their spinal muscles as forcefully, whereas gluteus maximus activity remained low in all groups because the tasks were unloaded.

Practical Take-Aways

* Hamstrings shorter than about 60 ° on the SLR "lock" the pelvis and make the lower back bend excessively, increasing spinal strain.
* Improving hamstring length shifts motion back toward the pelvis, reducing demand on lumbar joints and muscles.
* Even small everyday bends-such as reaching for an object on a chair-follow the same pattern, so stretching benefits daily life, not just sports performance.
* Patients and families can adopt simple hamstring-stretch routines; clinicians should consider targeted flexibility training whenever SLR is 60 ° or below before progressing to heavy lifting or core-stability programs.

Limitations The study involved healthy young adults and measured only unloaded forward bending. Outcomes may differ in older individuals, manual laborers, or tasks that involve twisting or weight. Long-term research is needed to confirm that stretching actually prevents low-back pain.

Bottom Line Flexible hamstrings let the pelvis and lower back "share the job." If your hamstrings are tight, your spine must work harder, which may invite discomfort or injury over time. A regular stretching program that brings SLR above roughly 60 ° can restore a healthier, more balanced bending pattern and help protect the lower back.

DETAILED DESCRIPTION:
This cross-sectional biomechanical study investigates how reduced hamstring flexibility alters sagittal lumbopelvic rhythm and trunk-hip muscle activation during forward bending. All procedures are completed in a single laboratory visit and do not involve any clinical intervention or longitudinal follow-up.

Study setting and oversight Testing is conducted in a university motion-analysis laboratory equipped with force-isolated flooring, adjustable height fixtures, and electromagnetic shielding. The protocol was approved by the Institutional Review Board of Sahmyook University (IRB #SYU-2025-03-033-002). Written informed consent is obtained before any study-related activity, and the identity of participants is coded to protect confidentiality.

Participant allocation and sample size

A priori power analysis (one-way ANOVA, effect size f = 0.55, α = 0.05, power = 0.80) indicated that at least 36 participants were required; 38 healthy adults were enrolled to offset potential attrition, and 37 completed the protocol. Participants are not assigned to treatment arms but are retrospectively stratified into three flexibility categories based on their dominant-limb straight-leg-raise (SLR) angle:

(1) ≤ 60° (short group), (2) 61-79° (moderate group), (3) ≥ 80° (long group). Eligibility criteria-including absence of low-back pain in the preceding six months-are recorded in a separate module.

Instrumentation and calibration

* Inertial-measurement units (IMUs; Xsens MTw Awinda, 60 Hz) are affixed to T12, S2, and the posterior thigh with double-sided tape and elastic wraps after a two-point static calibration that aligns sensor axes with anatomical reference frames.
* Surface electromyography (EMG; Delsys Trigno, 1 000 Hz) records bilateral erector spinae at L3, multifidus at L5, biceps femoris long head, and gluteus maximus. Skin is shaved, abraded, and cleaned with 70 % alcohol; electrode pairs are placed parallel to muscle fibers following SENIAM guidelines.
* Maximal voluntary contractions (MVCs) for each muscle are collected for normalisation. All raw data are synchronised via a hardware trigger and stored in a de-identified repository.

Experimental tasks

After warm-up, participants perform two tasks in random order, three trials each, barefoot and with knees extended:

1. a full-range forward bend from upright to maximum comfortable flexion and return, and
2. a partial bend from upright to the point where fingertips touch the patella and return.

A metronome (80 beats · min-¹) standardises angular velocity. Verbal instructions avoid coaching specific pelvic or lumbar strategies.

Primary technical outcomes Sagittal lumbar and pelvic angles are derived from IMU quaternions and filtered with a fourth-order Butterworth filter (6 Hz). The Relative Contribution Index (RCI) is calculated as the percentage of total trunk excursion attributable to the lumbar spine, sampled at 10 % increments of the flexion and extension phases. Higher RCI indicates greater lumbar-dominant motion.

Secondary outcomes EMG envelopes are obtained via 20-450 Hz band-pass filtering, full-wave rectification, and 50 ms moving RMS smoothing, then normalised to MVC. Variables include phase-specific RMS amplitude, median-frequency shift (fatigue index), and onset latency relative to movement initiation (5° pelvic tilt threshold).

Quality assurance and data integrity A detailed standard-operating-procedure manual governs sensor placement, calibration, and data extraction. Two investigators independently inspect raw signals for artefacts such as sensor dropout, cable motion (EMG), or excessive noise (> 2 SD from baseline). Automated scripts perform range and consistency checks (e.g., lumbar angle cannot exceed 90°; EMG RMS must be below 100 % MVC in unloaded tasks). Raw and processed files are archived on an encrypted server with automated daily backup.

Source-data verification is performed on 15 % of records by an auditor who cross-checks digital files against paper consent and data-capture sheets. A project-level data dictionary (CSV format) defines every variable, its unit, permissible range, and coding scheme. Version-controlled MATLAB and Python scripts are maintained in a private Git repository, and changes trigger a checksum comparison to detect unintended alterations.

Plan for missing or unusable data Trials with sensor artefact, loss of synchrony, or premature task termination are repeated once immediately; if unusable, they are marked "missing." If < 10 % of RCI values are missing, single-imputation using predictive mean matching is applied; otherwise, the participant is excluded from that analysis. EMG values with motion artefact are processed by wavelet-based denoising; segments that remain unusable are set to missing and handled as above.

Statistical analysis The primary hypothesis (hamstring flexibility influences RCI) is tested with one-way ANOVA, followed by Bonferroni-corrected pairwise comparisons. Phase-specific differences are explored with mixed-effects models (fixed = group × phase, random = subject). Pearson or Spearman correlations (based on Shapiro-Wilk normality) quantify relations between SLR angle and continuous RCI or EMG variables. Significance is set at p < 0.05; effect sizes are reported as partial η² or r. Statistical analyses are performed in R (v4.3.2) with the "lme4" and "effectsize" packages.

Safety monitoring and adverse-event reporting The biomechanical tasks are low-risk; however, any adverse sensation (e.g., back discomfort) prompts immediate cessation and optional referral to on-campus physical-therapy services. Adverse events are documented in the electronic case-report form and reviewed weekly by the principal investigator; serious adverse events would be reported to the IRB within 24 hours, although none are anticipated.

Patient-registry considerations This investigation is not a patient registry; therefore, external certification, on-site audits, and participant-year calculations do not apply. Should future registry expansion occur, the quality-assurance framework described above provides the foundation for broader surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults without musculoskeletal or neurological impairments
* Individuals without lumbar spine and lower limb disorders
* Participants who provided voluntary written informed consent

Exclusion Criteria:

* History of lumbar surgery or significant trauma
* Presence of acute or chronic pain conditions in lumbar or hip regions
* Neurological or orthopedic disorders affecting lumbar and hip functions
* Pregnancy
* Individuals unable to perform the required physical activities safely

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthy young adults aged 18 - 40 years. Participants will be recruited from the local community and university settings. Individuals included are those without any known musculoskeletal or neurological impairments, specifically with no history of lumbar or lower limb disorders, and who voluntarily agree to participate after providing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Lumbar Relative Contribution Index (RCI) During Full-Range Forward Bend | Single assessment session (one day)
  Sagittal-plane RCI is defined as the percentage of total trunk excursion attributable to lumbar-spine motion while participants bend forward from upright to maximal comfortable flexion and return. Higher values indicate greater lumbar dominance. Mean RCI will be compared across three hamstring-flexibility groups (SLR ≤ 60°, 61-79°, ≥ 80°).
Lumbar Relative Contribution Index (RCI) During Partial Forward Bend | Single laboratory visit; data captured during a ~15-minute test session for each participant.
  The sagittal-plane RCI is defined as the percentage of total trunk-flexion excursion attributable to lumbar-spine motion while the participant bends forward only until the fingertips touch the patella and then returns to upright. IMU data (T12, S2) are filtered at 6 Hz and processed to compute lumbar and pelvic angles; RCI is sampled at 10 % increments of the flexion and extension phases. Mean RCI values will be compared across three hamstring-flexibility groups (SLR ≤ 60°, 61-79°, ≥ 80°).

SECONDARY OUTCOMES:
Mean Normalised RMS EMG Amplitude of Lumbar Erector Spinae During First Half of Full-Range Forward Bend | Single laboratory visit; data captured during a ~15-minute test session for each participant.
  Surface EMG signals are recorded bilaterally from the L3-level erector-spinae muscles (Delsys Trigno, 1 000 Hz). Signals are band-pass filtered (20-450 Hz), full-wave rectified, and smoothed with a 50 ms moving RMS window, then normalised to each participant's maximal voluntary contraction (%MVC). The outcome is the average %MVC amplitude measured during the first 50 % of the flexion phase of a full-range forward bend. Group differences between hamstring-flexibility strata will be analysed using one-way ANOVA followed by Bonferroni post-hoc tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahmyook University, Seoul, Nowon-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided